CLINICAL TRIAL: NCT07274475
Title: Exploring Alternative Approaches to Harm Reduction and Cessation for Treatment-Resistant Tobacco Dependence
Brief Title: Smoking Harm Reduction Using E-cigarettes and Cytisine
Acronym: SHRECC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Laurie Zawertailo, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/040; 2425-HQ-000023 (Other Grant/Funding Number: Health Canada)
Record Dates: First submitted 2025-05-29; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Smoking; Harm Reduction; Nicotine
Keywords: Cytisine; E-cigarettes; Smoking cessation; treatment-resistant; Addiction; Clinical intervention
MeSH Terms: conditions — Tobacco Smoking; Harm Reduction; Vaping; Smoking Cessation; Behavior, Addictive | interventions — cytisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cytisine group (Active Comparator): Participants treated with Cytisine for smoking cessation
  Interventions: Dietary Supplement: Cytisine
- E-cigarette group (Active Comparator): Participants treated with E-cigarettes for smoking cessation
  Interventions: Device: E-cigarette e-liquid

INTERVENTIONS:
Device: E-cigarette e-liquid — E-cigarette used as a smoking cessation intervention
  Arms: E-cigarette group
Dietary Supplement: Cytisine — Cytisine used as a smoking cessation intervention
  Arms: Cytisine group

SUMMARY:
Smoking remains the leading cause of preventable death globally, with high prevalence in disadvantaged populations despite access to free nicotine replacement therapy (NRT) and counseling through Ontario's STOP Program. This study aims to evaluate the acceptability, feasibility, and comparative effectiveness of e-cigarettes and cytisine as harm-reduction tools for individuals who continue to smoke despite standard treatments. Over four years, 6,000 STOP participants who smoke ≥5 cigarettes daily at six months post-treatment will be randomized to receive either an e-cigarette starter kit or a 28-day cytisine supply. Data will be collected via REDCap and include biomarkers (NNAL, PAH), self-reported smoking behavior, nicotine dependence, and quality of life. Statistical analyses will assess changes and compare outcomes between groups. Results will inform public health strategies and enhance equitable cessation support for underserved populations.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to comply with all study procedures, for the full duration of the study period (12 months);
2. Age 18 years or older;
3. Currently smoking 5 or more cigarettes daily; and
4. Must have regular access to a phone and email to receive study communications and complete study monitoring.

Exclusion Criteria:

1. Individuals who smoke only occasionally or have quit smoking prior to the 6-month follow-up;
2. Daily or almost daily users of e-cigarettes for the past 30 days;
3. Presence of medical or psychiatric conditions that may interfere with safe participation or compliance with the study protocol, including severe cardiovascular disorders, renal impairment or respiratory conditions;
4. Known allergy or hypersensitivity to any components of the e-cigarettes, e-liquids, or cytisine;
5. Pregnant or breastfeeding, or planning to become pregnant within the next 12 months; or
6. Current use of pharmacological smoking cessation aids or participation in other smoking cessation clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Voucher redemption rates as measures of feasibility for e-cigarettes and cytisine | From enrollment to the 12-month follow-up
  To test the feasibility of e-cigarettes and cytisine as alternatives to standard evidence-based treatment in a group of individuals who were unable to quit using standard evidence-based treatment of NRT and counselling.

SECONDARY OUTCOMES:
Effectiveness of e-cigarettes and cytisine for smoking cessation measured by change in cigarettes per day | From enrollment to the 12-month follow-up
  The objective is to compare the effectiveness of e-cigarettes and cytisine. The main effectiveness outcome is change from baseline in cigarettes per day (CPD) at end of treatment. Researchers will dichotomize this variable to assess the proportion of participants in each group that achieve ≥ 50% reduction in CPD.

IPD SHARING:
Plan to Share IPD: No